CLINICAL TRIAL: NCT06212154
Title: The Safety and Efficacy of ThisCART19A for Relapsed/Refractory Autoimmune Hemolytic Anemia Patients After Receiving Three or More Lines of Therapy.
Brief Title: CAR-T for Autoimmune Hemolytic Anemia Patients Who Have Failed Three or More Lines of Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Suzhou Fundamenta Therapeutics (Unknown)
Responsible Party: Principal Investigator, Jun Shi, Director of Regenerative Medicine Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT400-025
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Autoimmune Hemolytic Anemia; CD19 CAR-T Cell Infusion
Keywords: ThisCART19A; Autoimmune Hemolytic Anemia; Relapsed/refractory after receiving three or more lines of therapy
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19A (Experimental): ThisCART19A comprises of allogeneic T-cells, which are genetically engineered to express chimeric antigen receptor (CAR) and targets cells expressing CD19.
  Interventions: Biological: ThisCART19A

INTERVENTIONS:
Biological: ThisCART19A — Participants will receive ThisCART19A cell infusion after preconditioning, and they need to be closely monitored for 28 days following CAR-T cell infusion.
  Other Names: Allogeneic CAR-T targeting CD19

SUMMARY:
To Evaluate the Safety and Efficacy of ThisCART19A for Relapsed/Refractory Autoimmune Hemolytic Anemia Patients After Receiving Three or More Lines of Therapy

DETAILED DESCRIPTION:
This is a phase 1, single-arm, open-label, dose-escalation and dose-expansion study. The main purpose is to evaluate the safety and tolerability, efficacy, pharmacokinetics and pharmacodynamics of ThisCART19A in patients with autoimmune hemolytic anemia who have failed ≥3 lines of therapy, which include glucocorticoids, rituximab, cyclophosphamide, azathioprine, fludarabine, cyclosporine, mycophenolate mofetil, BTK inhibitors, splenectomy, etc. Participants will receive ThisCART19A cell infusion after preconditioning, and they need to be closely monitored for 28 days following CAR-T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or subject's legal personal representative fully understand and voluntarily sign informed consent forms.
* Male or female age ≥ 12 years.
* ECOG performance status ≤2.
* Diagnosis of warm antibody hemolytic anemia (AIHA), cold AIHA, mixed AIHA or Evans syndrome.
* Hemoglobin<100g/L.
* Failure or intolerance to at least 3 lines of therapy, including glucocorticoids, rituximab, cyclophosphamide, azathioprine, fludarabine, cyclosporine, mycophenolate mofetil, Bruton's tyrosine kinase inhibitors, splenectomy.
* Laboratory tests of adequate organ function: Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×ULN; Creatinine clearance (CrCl) (Cockcroft-Gault formula) ≥40ml/min; Absolute neutrophil count (ANC) ≥1.0×10^9/L (growth factors such as granulocyte colony-stimulating factor [G-CSF] were not received within 7 days before the screening period); Left ventricular ejection fraction (LVEF) ≥45%; Blood oxygen saturation (SpO2) ≥92%.
* Subjects of childbearing potential will be required to follow contraception requirements from the time of enrollment until the end of the 6-month safety follow-up period. Female subjects of childbearing potential must have a negative Serum HCG test within 7 days before enrollment and not in the lactation period.

Exclusion Criteria:

* Clear diagnosis of lymphoproliferative tumor.
* The platelet count in peripheral blood during the screening period is <20×10^9/L.
* Have a history of severe drug allergy or allergic constitution.
* Have a history of any of the following diseases: craniocerebral trauma, consciousness disorder, epilepsy, cerebrovascular ischemia, cerebrovascular, and hemorrhagic diseases within 6 months before enrollment.
* Have any of the following serious cardiovascular diseases: myocardial infarction within 6 months before enrollment, cardiac angioplasty or stent implantation); Unstable angina; Severe cardiac arrhythmias; History of severe nonischemic cardiomyopathy; Congestive heart failure (New York Heart Association [NYHA] Class III or IV)).
* Have malignant tumors within 5 years before enrollment, unless any of the following conditions: fully treated cervical carcinoma in situ, fully treated basal cell or squamous epithelial cell skin cancer, localized prostate cancer after radical mastectomy, breast ductal carcinoma in situ after radical mastectomy, Carcinoma in situ in other locations one year after radical resection, and these diseases have no evidence of relapse.
* Subjects with any serious active fungal, bacterial, viral, tuberculosis or other infections, including active hepatitis B (defined as serum HBV-DNA ≥ 2000 IU/mL), active hepatitis C virus (Hepatitis C virus (HCV) infection, human immunodeficiency virus (HIV) antibody-positive or active syphilis patients, etc. Subjects whose HBV-DNA < 2000 IU/mL can be included on the condition that they receive antiviral drugs and monitor the related indicators during the study.
* Have mental illness and severe cognitive impairment.
* Have a history of live attenuated vaccines within 4 weeks before enrollment.
* Subjects considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of treatment-emergent adverse events | Within 6 months
Maximal Tolerable Dose(MTD) | Up to 28 days after infusion
  MTD is classified by the NCI CTCAE V5.0

SECONDARY OUTCOMES:
Best response rate (BOR) of each dose group | Within 12 weeks after infusion
  BOR is determined as the most favorable response observed after cell infusion, until either disease relapse or the completion of a specified observation period.
Objective response rate (ORR) | Within 4 weeks after infusion
  Percentage of patients with hematological response
Time to response (TTR) | Within 6 months
  TTR is defined as the duration from cell infusion to the achievement of a hematological response

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China